CLINICAL TRIAL: NCT01479556
Title: Assessment of Pregabalin Efficacy for the Treatment and Prevention of At-level Non-evoked and Evoked Spinal Cord Injury Neuropathic Pain
Brief Title: Pregabalin for the Treatment and Prevention of Spinal Cord Injury Neuropathic Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Julian Taylor Green (Other)
Responsible Party: Sponsor-Investigator, Julian Taylor Green, Dr. Julian Taylor Green, Hospital Nacional de Parapléjicos de Toledo
Organization: Hospital Nacional de Parapléjicos de Toledo (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HNP-02-2011; 2011-000915-14 (EudraCT Number)
Record Dates: First submitted 2011-11-17; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Neuropathic Pain; Spinal Cord Injuries
Keywords: Pregabalin; Neuropathic pain; At-level neuropathic pain; Non-evoked neuropathic pain; Evoked neuropathic pain; Sub-acute spinal cord injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Study subjects wil be randomized to the Placebo arm following a stratification procedure based on AIS scale (A-E), neurological level of injury (cervical or thoracic), and presence of at-level neuropathic pain before or after 3 months from the time of spinal cord injury.
  Interventions: Drug: Placebo
- Pregabalin (Active Comparator): Study subjects wil be randomized to the Pregabalin arm following a stratification procedure based on AIS scale (A-E), neurological level of injury (cervical or thoracic), and presence of at-level neuropathic pain before or after 3 months from the time of spinal cord injury.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin Alpha2-delta calcium channel blocker. 150mg BID p.o.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — 150mg BID p.o.
  Arms: Placebo

SUMMARY:
This study is a phase IV clinical trial with the objective of evaluating whether pain relief associated with pregabalin for at-level non-evoked and evoked neuropathic pain is more efficient during the early rather than late subacute phase of spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Comprehension of clinical trial and signed informed consent before initiation.
* Male or female adults, age 18 to 70.
* Clinical history of neuropathic pain secondary to SCI
* Patients with an AIS of A, B, C or D according to the American Spinal Cord Injury Association (ASIA) Impairment Scale.
* Persistent neuropathic pain from 1 month up to 6 months after spinal cord injury.
* Non-evoked at-level pain with ≥ 2 intensity measured with the numerical rating scale (0-10).
* Non-evoked/evoked at-level pain corresponding to the area of sensory alteration, and within the three dermatomes below the neurological level of the spinal cord injury.
* Formal acceptance of disponibility for all programmed clinical trial visits and other protocol requisites.
* Females of child bearing age must demonstrate a negative pregnancy test (performed on screening and subsequent follow up visits) and use a reliable birth control method including abstinence of sexual activity throughout the duration of the study and for at last 28 days after termination of the clinical trial.

Exclusion Criteria:

* Previous or actual use of gabapentin.
* Creatinine clearance level <60 ml/min.
* Neuropathic pain unrelated to spinal cord injury.
* Lactose intolerance, Lapp lactase insufficiency or glucose malabsorption
* Platelet count < 100x103/µl.
* White blood cell count <2.5 x103/µl.
* Neutrophil count <1.5 x103/µl.
* Planned surgery during the clinical trial.
* Patients with peripheral neuropathic pain.
* Previous history of malignant melanoma.
* History of malignant tumors, except for in situ uterine cervix carcinoma, in situ basocellular or spinocellular cutaneous carcinomas, superficial bladder tumors (Ta and Tis) with a complete treatment response up to 10 years. Patients with history of lymphoma or breast cancer will be allowed to participate in the trial if a complete treatment response has been observed up to 20 years.
* Chronic or active infection requiring a systemic therapy, chronic kidney infections, chronic lung infections with bronchiectasias, Mycobacterium tuberculosis infection, active Hepatitis B or C. Diagnosis of latent TB confection should be performed according to the local guidelines.
* Severe heart diseases such as unstable angina, cardiopathy during the first 6 months after a myocardial infarction, grade III or IV of the New York Heart Association scale for congestive heart failure.
* Unknown kidney, liver, gastrointestinal, endocrine, lung, hematological, neurological or psychiatric comorbidities.
* Subjects administered with an experimental or non-commercial drug during the 4 weeks prior to the trial.
* Patients participating in other clinical studies.
* Patients that are not competent for completing required tasks (eg. alcohol or drug related problems or psychiatric disorders).
* Subjects unable to be examined with radiological MRI exploration due to contraindications.
* Pregnancy or breastfeeding.
* Any other patient condition that is deemed unsuitable for subject inclusion in the trial according to the research team.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-05 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Daily at-level non-evoked pain intensity measured with the numerical rating scale (0-10) expressed as the mean 7-day pain intensity

SECONDARY OUTCOMES:
Weekly below-level non-evoked pain intensity measured with the numerical rating scale (0-10)
Weekly evaluation of at-level neuropathic pain symptoms using the "Neuropathic Pain Symptoms Inventory" (NPSI)
Weekly evaluation of at-level neuropathic pain intensity and interference using the "Brief Pain Inventory" (BPI)
Weekly evaluation of the change in at-level non-evoked neuropathic pain using the "Patient Global Impression Change" (PGIC)
Weekly evaluation of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS)
Weekly evaluation of spasm frequency below the spinal cord injury using the Penn questionnaire
Measurement of the amplitude of cold and heat sensory evoked potentials (Cz-Fz) studied above (C4) and at-level of the SCI
Serum TNF-R1 level
Weekly at-level non-evoked pain intensity measured with the numerical rating scale (0-10) 28 days after the termination of the clinical trial
Number of Paracetamol tablets used as rescue medication during the week
Prevalence and type of adverse events in patients treated with pregabalin
Unblinding testing: patient and investigator will be asked for the treatment they think to have received. Reasons for their judgement (efficacy and safety) will also be asked.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nacional de Parapléjicos de Toledo, Toledo, Toledo, Spain